CLINICAL TRIAL: NCT03562832
Title: Phase II, Open Label Clinical Study to Investigate Anti-tumour Effect and Tolerability of the PARP Inhibitor 2X-121 in Patients With Metastatic Breast Cancer Selected by the 2X-121 DRP
Brief Title: Investigation of Anti-tumour Effect and Tolerability of the PARP Inhibitor 2X-121 in Patients With Metastatic Breast Cancer Selected by the 2X-121 DRP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allarity Therapeutics (Industry)
Collaborators: Smerud Medical Research International AS (Other); Danish Breast Cancer Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OV-121; SMR-3475 (Other: Smerud Medical Research International)
Record Dates: First submitted 2018-04-26; First posted 2018-06-20 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Breast Cancer
Keywords: PARP inhibitor; Drug Response Prediction (DRP); Tankyrase 1/2 inhibitor; mRNA biomarker
MeSH Terms: conditions — Breast Neoplasms | interventions — stenoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PARP inhibitor 2X-121 (Experimental): 600 mg PARP inhibitor 2X-121 as single daily oral agent in mBC patients
  Interventions: Drug: PARP inhibitor 2X-121

INTERVENTIONS:
Drug: PARP inhibitor 2X-121 — 600 mg PARP inhibitor 2X-121 as single daily oral agent in mBC patients

SUMMARY:
2X-121 is a small molecule targeted inhibitor of Poly ADP ribose polymerase (PARP), a key enzyme involved in DNA damage repair in cancer cells. The PARP inhibitor demonstrated clinical activity in a prior Phase 1 study in a number of solid tumors. 2X-121 has a novel dual-inhibitory action against both PARP 1/2 and Tankyrase 1/2. The molecule is also active in P-glycoprotein expressing cells, suggesting it may overcome some of the PARP inhibitor resistance.

The Phase 2 study is using 2x-121 DRP® biomarker in metastatic breast cancer patients to identify patients likely to respond to and benefit from treatment with 2X-121.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Age 18 years or older.
* Histologically or cytological documented mBC (independent of hormone receptor, HER2 status and BRCA1 or 2 status) relapsed in 2 or more different prior therapies.
* Measurable disease by CT scan or MRI.
* With a drug response prediction (DRP) for 2X-121 with an outcome measured as being in the upper 20% likelihood of response.
* Prior chemotherapy or hormone therapy for metastatic breast cancer is allowed.
* Performance status of ECOG <= 1
* Recovered to Grade 1 or less from prior surgery or from acute toxicities of prior radiotherapy, or from treatment with cytotoxic, hormonal or biologic agents).
* >= 2 weeks must have elapsed since any prior surgery or therapy with G-CSF and GM-CSF.
* Patients with intracranial disease must be on stable or decreased level of steroid therapy (e.g. dexamethasone) for at least 7 days prior to baseline MRI. Non-enzymatic inducing ant-epileptic drugs are allowed.
* Adequate conditions as evidenced by the following clinical laboratory values:

  * Absolute neutrophils count (ANC) >= 1.5 x 10E9/L
  * Haemoglobin is at least 4.6 mmol/L
  * Platelets >= 100 x 10E9 /L
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 x ULN*
  * Serum bilirubin <= 1.5 ULN
  * Alkaline phosphatase <= 2.5 x ULN*
  * Creatinine <= 1.5 ULN
  * Blood urea within normal limits
  * Creatinine clearance within normal limits. *In case of known liver metastases with ALT and AST <= 5 x ULN and/or alkaline phosphatase <= 5 x ULN. Patients who do not conform to the transaminase and/or alkaline phosphatase inclusion criteria, but who by the PI are considered in good PS and otherwise eligible for inclusion, and where the transaminase and/or alkaline phosphatase levels are considered elevated due to other reasons than deteriorated lever capacity, may be considered for inclusion based on conferred agreement between PI and sponsor.
* Life expectancy equal or longer than 3 months.
* Sexually active females of child-producing potential must use adequate contraception (oral contraceptives, intrauterine device or barrier method of contraception) for the study duration and at least six months afterwards.

Exclusion Criteria:

* - Concurrent chemotherapy, radiotherapy, hormonal therapy, or other investigational drug except non-disease related conditions (e.g. insulin for diabetes) during study period.
* Other malignancy with exception of curative treated non-melanoma skin cancer or cervical carcinoma in situ within 5 years prior to entering the study.
* Previous treatment with PARP inhibitors
* Any active infection requiring parenteral or oral antibiotic treatment.
* Has known HIV positivity.
* Has known active hepatitis B or C.
* Has clinical significant (i.e. active) cardiovascular disease:

  * Stroke within <= 6 months prior to day 1
  * Transient ischemic attach (TIA) within <= 6 months prior to day 1
  * Myocardial infarction within <= 6 months prior to day 1
  * Unstable angina
  * New York Hart Association (NYHA) Grade II or greater congestive heart failure (CHF)
  * Serious cardiac arrhythmia requiring medication
* Mental status is not fit for clinical study or CNS disease including symptomatic epilepsy.
* Other medications or conditions, including surgery, that in the Investigator's opinion would contraindicate study participation of safety reasons or interfere with the interpretation of study results
* Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the bioavailability of 2X-121.
* Requiring immediate palliative treatment of any kind including surgery and/or radiotherapy.
* Female patients who are pregnant or breast-feeding (pregnancy test with a positive result before study entry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Anti-tumour efficacy after treatment with 600 mg 2X-121 as single oral agent in a 21-days cycle in mBC patients selected by the 2X-121 DRP | one year
  Overall tumor response according to RECIST

SECONDARY OUTCOMES:
Progression free survival (PFS) after administration of 2X-121 in patients with mBC | one year
  Timespan
Duration of objective response after administration of 2X-121 in patients with mBC | one year
  Timespan
Overall survival (OS) after administration of 2X-121 in patients with mBC | one year
  Timespan
Performance status (ECOG) | one year
  To evaluate change in patient performance status by ECOG (Eastern Cooperative Oncology Group) Performance Status by a 6-step classification system
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | one year
  Adverse Events as assessed by CTCAE v4. to evaluate safety profile after administration of 2X-121 in patients with mBC

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Herlev and Gentofte Hospital, Herlev Ringvej 75, DK-2730 Herlev, Herlev
  - Vejle Sygehus, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Official Homepage of Sponsor — http://www.oncologyventure.com